CLINICAL TRIAL: NCT00426023
Title: Multicenter, Randomised, Double Masked, Controlled Studies on the Efficacy of Cyclosporine Eye Drop Treatment in Preventing Vernal Keratoconjunctivitis (VKC) Relapses and in Treating the Acute Phase.
Brief Title: Cyclosporin A Eye Drop Treatment in Vernal Keratoconjunctivitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Campus Bio-Medico University (Other)
Collaborators: University of Genova (Other); University of Padova (Other)
Responsible Party: Alessandro Lambiase, University of Rome Campus Bio-Medico
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: eudract 2006-003689-32; FARM5YZTZW; ALMA1
Record Dates: First submitted 2007-01-23; First posted 2007-01-24 (Estimated); Last update posted 2009-01-28 (Estimated); Status verified 2009-01

CONDITIONS: Vernal Keratoconjunctivitis
Keywords: Vernal keratoconjunctivitis; Cyclosporine; Children; Clinical trial
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — Ketotifen; Ophthalmic Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental): this group of patients is treated with the experimental drug (Cyclosporine A 0,05% eye drops) 2 times daily
  Interventions: Drug: Cyclosporine A 0,05% eye drop
- 2 (Active Comparator)
  Interventions: Drug: ketotifen fumarate 0.025% eye drops

INTERVENTIONS:
Drug: Cyclosporine A 0,05% eye drop — Cyclosporine A 0.05% eye drops will be administered 2 times daily for six months in the first year of the study and in the second year of the study in a cross-over manner(from March to September)
  Other Names: NOVA22007
  Arms: 1
Drug: ketotifen fumarate 0.025% eye drops — ketotifen fumarate 0.025% eye drops 2 times daily for 6 months in the first year of the study (from March to September) and 6 months in the same period in the second year of the study in cross over manner.
  Other Names: Zaditen collirio monodose
  Arms: 2

SUMMARY:
This interventional study aims to evaluate the efficacy of Cyclosporine eye drop treatment in preventing relapses of Vernal Keratoconjunctivitis (VKC) and in treating the acute phases of the disease.

DETAILED DESCRIPTION:
Vernal keratoconjunctivitis (VKC) is a severe allergic disease, characterised by chronic ocular surface inflammation with seasonal relapses. Active phases of VKC require treatment with topical steroids to control inflammation and corneal damage that may lead to impairment of visual function and severe ocular discomfort. To date, safe and effective therapies in preventing relapses and controlling active phases of VKC are not available. Few controlled trials have used topical Cyclosporine A (CsA) for the treatment of VKC. The present multicenter, double-masked, randomised, controlled clinical trial will allow to obtain further data on the safety and efficacy of topical treatment with Cyclosporine in patients affected by VKC. Moreover, this study will evaluate the efficacy of topical CsA in both preventing the relapses of VKC and controlling the active phases of the disease. It is important to highlight that Cyclosporine eye drops are not currently commercially available in Italy and must be custom-made by specialized pharmacies. As VKC mostly affects young patients, it influences their daily life and their social interactions. Moreover, the severe signs and symptoms of the disease result in frequent ophthalmologic controls, influencing school activities of children and working days for their parents with a relevant economic cost for the National Health System.

Comparisons: Efficacy of Cyclosporine A 0.05% eye-drops in preventing VKC relapses compared to standard antiallergic (Ketotifen fumarate 0.025% eye-drops) treatment, and efficacy of Cyclosporine A 0.1% eye-drops in controlling acute phases compared to antiinflammatory (Desametasone 0.15% eye drops) treatments.

ELIGIBILITY:
Inclusion Criteria:

* Patients affected by VKC will be enrolled by the three Centres involved in the project
* Diagnosis of VKC will be performed on the basis of personal and family history of systemic allergic diseases, clinical examination (presence of conjunctival tarsal and/or limbal papillae) and presence of eosinophils in the conjunctival scraping

Exclusion Criteria:

* Contact lens wearers
* Patients affected by other ocular diseases
* Patients subjected to ocular surgery in the preceding 6 months
* Patients under eye drop or systemic treatments for other diseases, or
* Patients enrolled in experimental trials in the preceding 6 months

Ages: 5 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Estimated)
Dates: Start 2007-02; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
To compare the number of relapses of ocular inflammation per year between cyclosporine and ketotifen treated groups. Relapses are defined as at least 100% increase of the sum of hyperemia, itching, Trantas dots and corneal involvement | 2 years

SECONDARY OUTCOMES:
Differences of specific symptoms and signs, of TSyS, TSS, Quick questionnaire subscales and biochemical and | 2 years
molecular parameters will be evaluated at baseline, after 1, 3 and 6 months of treatment and after 1 month of treatment discontinuation | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: alessandro lambiase, MD, Principal Investigator — University of Rome Campus Bio-Medico
Locations (3):
- Italy (3):
  - University of Rome Campus Bio-Medico, Rome, Rome
  - University of Genova, Genova
  - University of Padua, Padua

REFERENCES:
- [Background] Bonini S, Bonini S, Lambiase A, Marchi S, Pasqualetti P, Zuccaro O, Rama P, Magrini L, Juhas T, Bucci MG. Vernal keratoconjunctivitis revisited: a case series of 195 patients with long-term followup. Ophthalmology. 2000 Jun;107(6):1157-63. doi: 10.1016/s0161-6420(00)00092-0. PMID 10857837
- [Background] Bonini S, Lambiase A, Sgrulletta R, Bonini S. Allergic chronic inflammation of the ocular surface in vernal keratoconjunctivitis. Curr Opin Allergy Clin Immunol. 2003 Oct;3(5):381-7. doi: 10.1097/00130832-200310000-00011. PMID 14501439
- [Background] Bonini S, Barney NP, Schiavone M, Centofanti M, Berruto A, Bonini S, Allansmith MR. Effectiveness of nedocromil sodium 2% eyedrops on clinical symptoms and tear fluid cytology of patients with vernal conjunctivitis. Eye (Lond). 1992;6 ( Pt 6):648-52. doi: 10.1038/eye.1992.139. PMID 1337745
- [Background] Bonini S, Micera A, Iovieno A, Lambiase A, Bonini S. Expression of Toll-like receptors in healthy and allergic conjunctiva. Ophthalmology. 2005 Sep;112(9):1528; discussion 1548-9. doi: 10.1016/j.ophtha.2005.04.009. PMID 16023216
- [Background] Mendicute J, Aranzasti C, Eder F, Ostolaza JI, Salaberria M. Topical cyclosporin A 2% in the treatment of vernal keratoconjunctivitis. Eye (Lond). 1997;11 ( Pt 1):75-8. doi: 10.1038/eye.1997.14. PMID 9246280
- [Background] Secchi AG, Tognon MS, Leonardi A. Topical use of cyclosporine in the treatment of vernal keratoconjunctivitis. Am J Ophthalmol. 1990 Dec 15;110(6):641-5. doi: 10.1016/s0002-9394(14)77061-8. PMID 2248328
- [Background] Gupta V, Sahu PK. Topical cyclosporin A in the management of vernal keratoconjunctivitis. Eye (Lond). 2001 Feb;15(Pt 1):39-41. doi: 10.1038/eye.2001.10. PMID 11318292
- [Background] BenEzra D, Pe'er J, Brodsky M, Cohen E. Cyclosporine eyedrops for the treatment of severe vernal keratoconjunctivitis. Am J Ophthalmol. 1986 Mar 15;101(3):278-82. doi: 10.1016/0002-9394(86)90819-6. PMID 3953723
- [Background] Leonardi A. Vernal keratoconjunctivitis: pathogenesis and treatment. Prog Retin Eye Res. 2002 May;21(3):319-39. doi: 10.1016/s1350-9462(02)00006-x. PMID 12052387